CLINICAL TRIAL: NCT02436239
Title: An Open-label Long-term Safety Study of Vilazodone in Pediatric Patients With Major Depressive Disorder
Brief Title: A Study of Vilazodone in Pediatric Patients With Major Depressive Disorder
Acronym: VLZ-MD-23
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VLZ-MD-23
Record Dates: First submitted 2015-04-28; First posted 2015-05-06 (Estimated); Results first posted 2019-09-11 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Vilazodone Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vilazodone (Experimental)
  Interventions: Drug: Vilazodone

INTERVENTIONS:
Drug: Vilazodone — Vilazodone tablets, once daily, oral administration
  Other Names: Viibryd

SUMMARY:
The purpose of this study is to evaluate the long-term safety and tolerability of vilazodone for the treatment of MDD in pediatric outpatients (7-17 years).

ELIGIBILITY:
Inclusion Criteria:

* Male or Female outpatients betw een 7-17 years of age
* Primary diagnosis of major depressive disorder (MDD)
* Children's Depression Rating Scale-Revised (CDRS-R) score of 40 or greater
* Clinical Global Impressions-Severity (CGI-S) score of 4 or greater

Exclusion Criteria:

* Current (past 3 months) principal Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision based diagnosis of an Axis I disorder other than MDD that is the primary focus of treatment (de novo patients only)
* History of suicidal behavior, or requires precaution against suicide
* Not generally healthy medical condition
* Seizure disorder

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 330 (Actual)
Dates: Start 2015-05-02 (Actual); Primary Completion 2018-07-23 (Actual); Study Completion 2018-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily McCusker, PhD, Study Director — Forest Research Institute, Inc., an affiliate of Allergan, plc
Locations (56):
- United States (54):
  - Alliance Clinical Research, Birmingham, Alabama
  - Harmonex Neuroscience Research, Dothan, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Woodland International Research Group, INC, Little Rock, Arkansas
  - CITrials - Bellflower, Bellflower, California
  - ATP Clinical Research, Costa Mesa, California
  - Behavioral Research Specialists, LLC, Glendale, California
  - PCSD - Feighner Research, San Diego, California
  - Pacific Clinical Research Medical Group, Hartford, Connecticut
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Palm Springs Research, LLC, Hialeah, Florida
  - IMIC Inc., Homestead, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Innovative Clinical Research, Inc., Lauderhill, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Institute for Advanced Medical Research, Alpharetta, Georgia
  - Atlantic Center for Medical Research, Atlanta, Georgia
  - Northwest Behavioral Research Center, Marietta, Georgia
  - Capstone Clinical Research, Libertyville, Illinois
  - Baber Research Group, Naperville, Illinois
  - Neuroscience Research Institute Inc., Oak Park, Illinois
  - Psychiatric Associates, Overland Park, Kansas
  - Lake Charles Clinical Trials, Lake Charles, Louisiana
  - Hugo W Moser Research Institute at Kennedy Krieger, Inc., Baltimore, Maryland
  - Pharmsite Research Inc., Baltimore, Maryland
  - NeuroScientific Insights, Rockville, Maryland
  - Baystate Medical Center, Springfield, Massachusetts
  - Adams Clinical Trials, LLC, Watertown, Massachusetts
  - Millennium Psychiatric Associates, Creve Coeur, Missouri
  - St. Charles Psychiatric Associates - Midwest Research Group, Saint Charles, Missouri
  - Erie County Medical Center/State University of New York of Buffalo Affiliate, Buffalo, New York
  - BioScience Research LLC, Mount Kisco, New York
  - Manhattan Behavioral Medicine, New York, New York
  - Finger Lakes Clinical research, Rochester, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - Haidar Almhana Nieding LLC, Avon Lake, Ohio
  - Neuro-Behavioral Clinical Research, Inc, Canton, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Psychiatr, Cleveland, Ohio
  - Ohio State Univ. Dept of Psychiatry, Columbus, Ohio
  - Professional Psychiatric Services, Mason, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Cutting Edge Research Group, Oklahoma City, Oklahoma
  - Research Strategies of Memphis LLC, Memphis, Tennessee
  - BioBehavioral Research of Austin, PC, Austin, Texas
  - UT Health Science Center at Houston, Houston, Texas
  - Houston Endoscopy and Research Ctr, Houston, Texas
  - Research Across America, Plano, Texas
  - Focus and Balance, San Antonio, Texas
  - Family Psychiatry of The Woodlands, The Woodlands, Texas
  - Ericksen Research and Development, Clinton, Utah
  - UVA Center for Psychopharmacology Research in Youth, Charlottesville, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - Core Clinical Research, Kirkland, Washington
- Canada (2):
  - Okanagan Clinical Trials Inc., Kelowna, British Columbia
  - Paediatric Sleep Research Inc, Toronto, Ontario

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients who completed lead-in study VLZ-MD-22 (NCT02372799) had already completed a down-taper period at the end of study VLZ-MD-22 and were not required to undergo a washout period in VLZ-MD-23. For de novo patients, the screening/washout period was generally 1 week prior to Baseline.
Groups:
- Placebo/Vilazodone: Participants who received placebo during the lead in study, VLZ-MD-22, were given vilazodone tablets once daily, oral administration.
- Vilazodone/Vilazodone: Participants who received vilazodone during the lead in study, VLZ-MD-22, were given vilazodone tablets once daily, oral administration.
- Fluoxetine/Vilazodone: Participants who received Fluoxetine during the lead in study, VLZ-MD-22, were given vilazodone tablets once daily, oral administration.
- De Novo/Vilazodone: Newly enrolled participants received vilazodone tablets once daily, oral administration.
Period: Open-Lable Treatment Period
Arm/Group | Placebo/Vilazodone | Vilazodone/Vilazodone | Fluoxetine/Vilazodone | De Novo/Vilazodone
Started | 122 | 131 | 65 | 12
Completed | 89 | 97 | 38 | 7
Not Completed | 33 | 34 | 27 | 5
Not completed — Adverse Event | 12 | 3 | 4 | 2
Not completed — Lack of Efficacy | 1 | 6 | 6 | 1
Not completed — Withdrawal by Subject | 10 | 15 | 9 | 0
Not completed — Lost to Follow-up | 4 | 2 | 4 | 1
Not completed — Protocol Violation | 0 | 1 | 1 | 0
Not completed — Noncompliance with Study Drug | 5 | 6 | 3 | 1
Not completed — Other Reason | 1 | 1 | 0 | 0
Period: Down-Taper Period
Arm/Group | Placebo/Vilazodone | Vilazodone/Vilazodone | Fluoxetine/Vilazodone | De Novo/Vilazodone
Started | 90 (Enrollment permitted for participants who had not completed previous open-label treatment period.) | 103 (Enrollment permitted for participants who had not completed previous open-label treatment period.) | 44 (Enrollment permitted for participants who had not completed previous open-label treatment period.) | 6 (One participant who completed the open-label treatment period did not enter the down-taper period.)
Completed | 86 | 99 | 43 | 4
Not Completed | 4 | 4 | 1 | 2
Not completed — Withdrawal by Subject | 4 | 4 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo/Vilazodone | Vilazodone/Vilazodone | Fluoxetine/Vilazodone | De Novo/Vilazodone | Total
Number analyzed (Participants) | 122 | 131 | 65 | 12 | 330
Age, Continuous [Mean (Standard Deviation); unit: Years] | 13.2 (2.9) | 13.3 (2.8) | 13.2 (2.8) | 13.0 (2.9) | 13.3 (2.9)
Age, Customized [Count of Participants; unit: Participants]
  Age 7-11 Years | 37 | 35 | 19 | 4 | 95
  Age 12-17 Years | 83 | 93 | 46 | 8 | 230
  Age 18 Years | 2 | 3 | 0 | 0 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 89 | 33 | 7 | 197
  Male | 54 | 42 | 32 | 5 | 133
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 16 | 8 | 2 | 42
  Not Hispanic or Latino | 106 | 115 | 57 | 10 | 288
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 5 | 1 | 1 | 0 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 0 | 0 | 2
  Black or African American | 32 | 40 | 20 | 1 | 93
  White | 82 | 84 | 42 | 11 | 219
  More than one race | 3 | 4 | 2 | 0 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] | 57.98 (23.54) | 62.67 (25.26) | 59.36 (18.93) | 60.34 (17.87) | 60.17 (23.26)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 22.73 (6.59) | 24.75 (7.96) | 23.30 (5.37) | 23.90 (6.20) | 23.69 (6.98)
CDRS-R total score [Mean (Standard Deviation); unit: units on a scale] — The Children's Depression Rating Scale-Revised (CDRS-R) total score ranges from 17 (minimal or no symptoms of depression) to 133 (indicative of depression) is a semi-structured, clinician-rated instrument designed for use with children and adolescents between the ages of 6 to 17 years of age and their caregivers. The CDRS-R evaluates the presence and severity of symptoms commonly associated with depression in childhood. Population: The CDRS-R total score is provided at baseline for the Intent to Treat study population, which comprises the 325 patients in the Safety Population who had a baseline and at least 1 postbaseline assessment of the CDRS-R total score.
  units on a scale
    number analyzed (Participants) | 121 | 130 | 63 | 11 | 325
    (all) | 55.7 (9.6) | 59.3 (9.5) | 57.8 (8.7) | 59.7 (9.1) | 58.4 (9.3)
CGI-S score [Mean (Standard Deviation); unit: units on a scale] — The Clinical Global Impressions-Severity (CGI-S) is a clinician-rated instrument used to rate the severity of the patient's current state of mental illness compared with the clinician's total experience with patients with major depressive disorder (MDD). The severity of the patient's MDD was rated on a scale from 1 to 7, with 1 indicating a normal state and 7 indicating a patient who is among the most extremely ill patients. Population: The CGI-S score is provided at baseline for the Intent to Treat study population, which comprises the 325 patients in the Safety Population who had a baseline and at least 1 postbaseline assessment of the CDRS-R total score.
  units on a scale
    number analyzed (Participants) | 121 | 130 | 63 | 11 | 325
    (all) | 4.6 (0.6) | 4.7 (0.7) | 4.6 (0.6) | 4.2 (0.4) | 4.6 (0.6)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants to Experience a Treatment Emergent Adverse Event (TEAE)
Description: The number of Participants who experienced a treatment emergent adverse events during the 27 week period from screening to the end of the open-label treatment period
Time Frame: Visit 1 (Week -1) to up to Visit 16 (Week 26)
Population: The Safety Population consisted of the 330 participants who took at least 1 dose of open-label investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo/Vilazodone | Vilazodone/Vilazodone | Fluoxetine/Vilazodone | De Novo/Vilazodone
Number analyzed (Participants) | 122 | 131 | 65 | 12
Participants | 90 | 89 | 48 | 10

2. Secondary Outcome: Change From Baseline in the CDRS-R Total Score
Description: The Children's Depression Rating Scale-Revised (CDRS-R) total score ranges from 17 (minimal or no symptoms of depression) to 133 (indicative of depression) is a semi-structured, clinician-rated instrument designed for use with children and adolescents between the ages of 6 to 17 years of age and their caregivers. The CDRS-R evaluates the presence and severity of symptoms commonly associated with depression in childhood.
Time Frame: Baseline (Week 0) to Week 26
Population: The Change From Baseline in the CDRS-R Total Score was assessed in the Intent to Treat study population, comprised of the 325 patients in the Safety Population who had a baseline and at least 1 postbaseline assessment of the CDRS-R total score.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo/Vilazodone | Vilazodone/Vilazodone | Fluoxetine/Vilazodone | De Novo/Vilazodone
Number analyzed (Participants) | 121 | 130 | 63 | 11
units on a scale | -29.2 (11.9) | -30.1 (12.2) | -29.4 (12.2) | -24.5 (10.3)

3. Secondary Outcome: Change From Baseline in the CGI-S Score
Description: The Clinical Global Impressions-Severity (CGI-S) is a clinician-rated instrument used to rate the severity of the patient's current state of mental illness compared with the clinician's total experience with patients with major depressive disorder (MDD). The severity of the patient's MDD was rated on a scale from 1 to 7, with 1 indicating a normal state and 7 indicating a patient who is among the most extremely ill patients.
Time Frame: Baseline (Week 0) to Week 26
Population: The CGI-S was assessed in the Intent to Treat study population, comprised of the 325 patients in the Safety Population who had a baseline and at least 1 postbaseline assessment of the CDRS-R total score.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo/Vilazodone | Vilazodone/Vilazodone | Fluoxetine/Vilazodone | De Novo/Vilazodone
Number analyzed (Participants) | 121 | 130 | 63 | 11
units on a scale | -2.5 (1.3) | -2.6 (1.4) | -2.5 (1.4) | -1.7 (1.2)

4. Secondary Outcome: Change From Baseline in Clinical Global Impressions-Improvement (CGI-I)
Description: The Clinical Global Impressions-Improvement is a clinician-rated instrument that was used to rate total improvement or worsening of mental illness, regardless of whether the Investigator considered it to be a result of treatment with the investigational product. The CGI-I was used to rate the patient's improvement on a scale from 1 to 7, with 1 indicating that the patient was very much improved (with a score of 4 indicating no change) and 7 indicating the patient was very much worse.
Time Frame: Baseline (Week 0) to Week 26
Population: The CGI-I was assessed in the Intent to Treat study population, comprised of the 325 patients in the Safety Population who had a baseline and at least 1 postbaseline assessment of the CDRS-R total score.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo/Vilazodone | Vilazodone/Vilazodone | Fluoxetine/Vilazodone | De Novo/Vilazodone
Number analyzed (Participants) | 121 | 130 | 63 | 11
units on a scale | 2.1 (1.2) | 2.0 (1.3) | 2.0 (1.2) | 2.2 (1.2)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for up to 28 weeks, which consists of the screening visit (1 week), the 26 week open label treatment period and during the 1 week down taper period.
Arm/Group | Placebo/Vilazodone | Vilazodone/Vilazodone | Fluoxetine/Vilazodone | De Novo/Vilazodone
All-Cause Mortality (participants affected / at risk) | 0/122 | 0/131 | 1/65 | 0/12
Serious Adverse Events (participants affected / at risk) | 6/122 | 0/131 | 1/65 | 0/12
Other Adverse Events (participants affected / at risk) | 79/122 | 81/131 | 41/65 | 10/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/Vilazodone (N=122) | Vilazodone/Vilazodone (N=131) | Fluoxetine/Vilazodone (N=65) | De Novo/Vilazodone (N=12)
Suicidal ideation (Psychiatric disorders) | 2 | 0 | 0 | 0
Abnormal behaviour (Psychiatric disorders) | 1 | 0 | 0 | 0
Aggression (Psychiatric disorders) | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0
Gun Shot Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/Vilazodone (N=122) | Vilazodone/Vilazodone (N=131) | Fluoxetine/Vilazodone (N=65) | De Novo/Vilazodone (N=12)
Ear Pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 2
Nausea (Gastrointestinal disorders) | 27 | 16 | 8 | 2
Vomiting (Gastrointestinal disorders) | 15 | 8 | 3 | 0
Abdominal pain upper (Gastrointestinal disorders) | 12 | 6 | 4 | 0
Nasopharyngitis (Infections and infestations) | 5 | 11 | 2 | 0
Gastroenteritis (Infections and infestations) | 6 | 3 | 3 | 1
Sinusitis (Infections and infestations) | 1 | 5 | 2 | 1
Weight increased (Investigations) | 7 | 15 | 4 | 1
Headache (Nervous system disorders) | 21 | 28 | 8 | 2
Dizziness (Nervous system disorders) | 3 | 9 | 4 | 0
Migraine (Nervous system disorders) | 3 | 3 | 1 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 2
Insomnia (Psychiatric disorders) | 13 | 11 | 2 | 0
Dysmenorrhea (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 3 | 0
Irritability (Psychiatric disorders) | 4 | 3 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 2 | 0 | 1
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data generated in this study are the property of the sponsor. An integrated clinical and statistical report will be prepared at the completion of the study. Publication of the results by the Investigator will be subject to mutual agreement between the Investigator and the sponsor and will follow sponsor's standard operating procedures on publications.

DOCUMENTS (2):
  • Study Protocol (2016-11-02): https://cdn.clinicaltrials.gov/large-docs/39/NCT02436239/Prot_000.pdf
  • Statistical Analysis Plan (2016-02-10): https://cdn.clinicaltrials.gov/large-docs/39/NCT02436239/SAP_001.pdf